CLINICAL TRIAL: NCT01301352
Title: The Efficacy and Safety of Gastric Feeding in Critically Ill Pediatric Patients Receiving Non-invasive Positive Pressure Ventilation: A Pilot Study
Brief Title: Feeding Children Nasogastrically Versus Nasojejunally While Receiving Noninvasive Positive Pressure Ventilation
Acronym: FeedNIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Allon Beck, Dr., McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 10-192-PED
Record Dates: First submitted 2011-02-22; First posted 2011-02-23 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Respiratory Insufficiency; Pneumonia, Aspiration; Nutrition Disorders
Keywords: Critical Care; Intubation, gastrointestinal; Child; Infant; Adolescent; Continuous positive airway pressure; Enteral Nutrition
MeSH Terms: conditions — Respiratory Insufficiency; Pneumonia, Aspiration; Nutrition Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nasojejunal feeding (control) (No Intervention)
- Nasogastric feeding (intervention) (Experimental)
  Interventions: Other: Route of feeding (nasogastric vs. nasojejunal)

INTERVENTIONS:
Other: Route of feeding (nasogastric vs. nasojejunal) — Safety and efficacy of feeding nasogastrically vs. nasojejunally while receiving noninvasive positive pressure ventilation
  Arms: Nasogastric feeding (intervention)

SUMMARY:
The investigators are studying whether it is safe and effective to provide enteral nutrition to critically ill children via the nasogastric route, as opposed to the nasojejunal route, while they are receiving noninvasive positive pressure ventilation.

DETAILED DESCRIPTION:
It has been our experience that the placement of post-pyloric tubes can be difficult, and that these tubes frequently become obstructed and are difficult to replace, resulting in lost caloric intake for the patient. The population where this is most relevant is children receiving Noninvasive Positive Pressure Ventilation (NPPV). NPPV has become increasingly popular in the Pediatric Intensive Care Unit (PICU) population, due to its perception as a safe and effective alternative to mechanical ventilation via an endotracheal tube. Historically, NPPV has been used in children with chronic respiratory insufficiency, but its application for acute respiratory compromise is increasing. It has been shown to be effective in disease states associated with hypoventilation, and is now also being applied to respiratory problems leading to decreased oxygenation. Infants and children receiving noninvasive ventilation for respiratory failure, which is often infectious in origin, have significant caloric needs. However, it is our practice not to allow gastric feeding in these patients due to the fear of gastric distension and vomiting, which carries a risk of aspiration.

There is no data available on the question of efficacy and safety of gastric feeding in critically-ill children supported by noninvasive ventilation. Given the ease of (re)placement, and the potential nutritional benefit of earlier feeding provided by gastric feeding, it seems clinically important to question the bias against this route of enteral nutrition in noninvasively ventilated patients. The investigators therefore propose a pilot randomized trial of gastric versus post-pyloric feeds in patients on NPPV.

ELIGIBILITY:
Inclusion Criteria:

* Age under 18 years old
* Acute respiratory failure as the indication for non-invasive ventilatory support
* Signed consent from parent or guardian
* Patients with a feeding tube in place who have not been fed in > 12 hours

Exclusion Criteria:

* Immediate postoperative cardiac surgery
* Chronic ventilatory support
* Admission diagnosis of aspiration pneumonia
* Known history of frequent aspiration (more than 2 previous admissions for this diagnosis)
* Contraindication to feeding tube placement (e.g. basal skull fracture)
* Imminent need for endotracheal intubation
* Percutaneous gastric tube in place
* History of Nissen fundoplication
* Contraindication to study nutritional formulas (e.g. galactosemia)
* Allergy to metoclopramide
* No signed consent from parent or guardian
* Continuous Positive Airway Pressure (CPAP) with or without pressure support administered via an endotracheal tube
* Corrected gestational age under 38 weeks
* Patients with a feeding tube in place who have been fed within the last 12 hours
* Patients with a feeding tube in place in whom the PICU staff do not wish to change the position of the feeding tube (i.e. do not agree to randomize the patient's feeding tube position)

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The percent goal enteral calories received while receiving NPPV | Daily up to 14 days
  Daily percent goal calories are recorded. Also total percent goal calories over entire NPPV course.

SECONDARY OUTCOMES:
The time required to achieve goal calories while on NPPV | Hours (estimated up to 48 hours)
The length of stay in ICU and in hospital | Days (estimated up to 14 and 28 days, respectively)
Episodes of clinically important gastric aspiration | Episodes (number - up to 1 per subject)

CONTACTS AND LOCATIONS:
Overall Officials: Pramod Puligandla, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal Children's Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Alberda C, Gramlich L, Jones N, Jeejeebhoy K, Day AG, Dhaliwal R, Heyland DK. The relationship between nutritional intake and clinical outcomes in critically ill patients: results of an international multicenter observational study. Intensive Care Med. 2009 Oct;35(10):1728-37. doi: 10.1007/s00134-009-1567-4. Epub 2009 Jul 2. PMID 19572118
- [Background] Antonelli M, Azoulay E, Bonten M, Chastre J, Citerio G, Conti G, De Backer D, Lemaire F, Gerlach H, Hedenstierna G, Joannidis M, Macrae D, Mancebo J, Maggiore SM, Mebazaa A, Preiser JC, Pugin J, Wernerman J, Zhang H. Year in review in Intensive Care Medicine 2009. Part III: mechanical ventilation, acute lung injury and respiratory distress syndrome, pediatrics, ethics, and miscellanea. Intensive Care Med. 2010 Apr;36(4):567-84. doi: 10.1007/s00134-010-1781-0. Epub 2010 Feb 23. No abstract available. PMID 20177660
- [Background] Barr J, Hecht M, Flavin KE, Khorana A, Gould MK. Outcomes in critically ill patients before and after the implementation of an evidence-based nutritional management protocol. Chest. 2004 Apr;125(4):1446-57. doi: 10.1378/chest.125.4.1446. PMID 15078758
- [Background] Binnekade JM, Tepaske R, Bruynzeel P, Mathus-Vliegen EM, de Hann RJ. Daily enteral feeding practice on the ICU: attainment of goals and interfering factors. Crit Care. 2005 Jun;9(3):R218-25. doi: 10.1186/cc3504. Epub 2005 Mar 22. PMID 15987393
- [Background] Braunschweig CL, Levy P, Sheean PM, Wang X. Enteral compared with parenteral nutrition: a meta-analysis. Am J Clin Nutr. 2001 Oct;74(4):534-42. doi: 10.1093/ajcn/74.4.534. PMID 11566654
- [Background] Cahill NE, Dhaliwal R, Day AG, Jiang X, Heyland DK. Nutrition therapy in the critical care setting: what is "best achievable" practice? An international multicenter observational study. Crit Care Med. 2010 Feb;38(2):395-401. doi: 10.1097/CCM.0b013e3181c0263d. PMID 19851094
- [Background] Casaer MP, Mesotten D, Schetz MR. Bench-to-bedside review: metabolism and nutrition. Crit Care. 2008;12(4):222. doi: 10.1186/cc6945. Epub 2008 Aug 19. PMID 18768091
- [Background] Essouri S, Durand P, Chevret L, Haas V, Perot C, Clement A, Devictor D, Fauroux B. Physiological effects of noninvasive positive ventilation during acute moderate hypercapnic respiratory insufficiency in children. Intensive Care Med. 2008 Dec;34(12):2248-55. doi: 10.1007/s00134-008-1202-9. Epub 2008 Aug 19. PMID 18712350
- [Background] Esteban A, Frutos-Vivar F, Ferguson ND, Arabi Y, Apezteguia C, Gonzalez M, Epstein SK, Hill NS, Nava S, Soares MA, D'Empaire G, Alia I, Anzueto A. Noninvasive positive-pressure ventilation for respiratory failure after extubation. N Engl J Med. 2004 Jun 10;350(24):2452-60. doi: 10.1056/NEJMoa032736. PMID 15190137
- [Background] Gramlich L, Kichian K, Pinilla J, Rodych NJ, Dhaliwal R, Heyland DK. Does enteral nutrition compared to parenteral nutrition result in better outcomes in critically ill adult patients? A systematic review of the literature. Nutrition. 2004 Oct;20(10):843-8. doi: 10.1016/j.nut.2004.06.003. PMID 15474870
- [Background] Greenough A. Role of ventilation in RSV disease: CPAP, ventilation, HFO, ECMO. Paediatr Respir Rev. 2009 Jun;10 Suppl 1:26-8. doi: 10.1016/S1526-0542(09)70012-0. PMID 19651398
- [Background] Griffiths RD. Is parenteral nutrition really that risky in the intensive care unit? Curr Opin Clin Nutr Metab Care. 2004 Mar;7(2):175-81. doi: 10.1097/00075197-200403000-00012. PMID 15075709
- [Background] Griffiths RD, Bongers T. Nutrition support for patients in the intensive care unit. Postgrad Med J. 2005 Oct;81(960):629-36. doi: 10.1136/pgmj.2005.033399. PMID 16210458
- [Background] Gurgueira GL, Leite HP, Taddei JA, de Carvalho WB. Outcomes in a pediatric intensive care unit before and after the implementation of a nutrition support team. JPEN J Parenter Enteral Nutr. 2005 May-Jun;29(3):176-85. doi: 10.1177/0148607105029003176. PMID 15837777
- [Background] Hadfield RJ, Sinclair DG, Houldsworth PE, Evans TW. Effects of enteral and parenteral nutrition on gut mucosal permeability in the critically ill. Am J Respir Crit Care Med. 1995 Nov;152(5 Pt 1):1545-8. doi: 10.1164/ajrccm.152.5.7582291.
- [Background] Hernandez G, Velasco N, Wainstein C, Castillo L, Bugedo G, Maiz A, Lopez F, Guzman S, Vargas C. Gut mucosal atrophy after a short enteral fasting period in critically ill patients. J Crit Care. 1999 Jun;14(2):73-7. doi: 10.1016/s0883-9441(99)90017-5. PMID 10382787
- [Background] Heyland DK, Cook DJ, Dodek PM. Prevention of ventilator-associated pneumonia: current practice in Canadian intensive care units. J Crit Care. 2002 Sep;17(3):161-7. doi: 10.1053/jcrc.2002.35814. PMID 12297991
- [Background] Heyland DK, Dhaliwal R, Drover JW, Gramlich L, Dodek P; Canadian Critical Care Clinical Practice Guidelines Committee. Canadian clinical practice guidelines for nutrition support in mechanically ventilated, critically ill adult patients. JPEN J Parenter Enteral Nutr. 2003 Sep-Oct;27(5):355-73. doi: 10.1177/0148607103027005355. PMID 12971736
- [Background] Heyland DK, Drover JW, MacDonald S, Novak F, Lam M. Effect of postpyloric feeding on gastroesophageal regurgitation and pulmonary microaspiration: results of a randomized controlled trial. Crit Care Med. 2001 Aug;29(8):1495-501. doi: 10.1097/00003246-200108000-00001. PMID 11505114
- [Background] Ho KM, Dobb GJ, Webb SA. A comparison of early gastric and post-pyloric feeding in critically ill patients: a meta-analysis. Intensive Care Med. 2006 May;32(5):639-49. doi: 10.1007/s00134-006-0128-3. Epub 2006 Mar 29. PMID 16570149
- [Background] Jabbar A, McClave SA. Pre-pyloric versus post-pyloric feeding. Clin Nutr. 2005 Oct;24(5):719-26. doi: 10.1016/j.clnu.2005.03.003. PMID 16143431
- [Background] Joshi G, Tobias JD. A five-year experience with the use of BiPAP in a pediatric intensive care unit population. J Intensive Care Med. 2007 Jan-Feb;22(1):38-43. doi: 10.1177/0885066606295221. PMID 17259567
- [Background] Kallet RH, Diaz JV. The physiologic effects of noninvasive ventilation. Respir Care. 2009 Jan;54(1):102-15. PMID 19111110
- [Background] Kawati R, Rubertsson S. Malpositioning of fine bore feeding tube: a serious complication. Acta Anaesthesiol Scand. 2005 Jan;49(1):58-61. doi: 10.1111/j.1399-6576.2005.00508.x. PMID 15675983
- [Background] Marik PE, Zaloga GP. Gastric versus post-pyloric feeding: a systematic review. Crit Care. 2003 Jun;7(3):R46-51. doi: 10.1186/cc2190. Epub 2003 May 6. PMID 12793890
- [Background] Mayordomo-Colunga J, Medina A, Rey C, Diaz JJ, Concha A, Los Arcos M, Menendez S. Predictive factors of non invasive ventilation failure in critically ill children: a prospective epidemiological study. Intensive Care Med. 2009 Mar;35(3):527-36. doi: 10.1007/s00134-008-1346-7. Epub 2008 Nov 4. PMID 18982307
- [Background] McClave SA, DeMeo MT, DeLegge MH, DiSario JA, Heyland DK, Maloney JP, Metheny NA, Moore FA, Scolapio JS, Spain DA, Zaloga GP. North American Summit on Aspiration in the Critically Ill Patient: consensus statement. JPEN J Parenter Enteral Nutr. 2002 Nov-Dec;26(6 Suppl):S80-5. doi: 10.1177/014860710202600613. PMID 12405628
- [Background] Meert KL, Daphtary KM, Metheny NA. Gastric vs small-bowel feeding in critically ill children receiving mechanical ventilation: a randomized controlled trial. Chest. 2004 Sep;126(3):872-8. doi: 10.1378/chest.126.3.872. PMID 15364769
- [Background] Metheny NA. Preventing respiratory complications of tube feedings: evidence-based practice. Am J Crit Care. 2006 Jul;15(4):360-9. PMID 16823013
- [Background] Montejo JC, Grau T, Acosta J, Ruiz-Santana S, Planas M, Garcia-De-Lorenzo A, Mesejo A, Cervera M, Sanchez-Alvarez C, Nunez-Ruiz R, Lopez-Martinez J; Nutritional and Metabolic Working Group of the Spanish Society of Intensive Care Medicine and Coronary Units. Multicenter, prospective, randomized, single-blind study comparing the efficacy and gastrointestinal complications of early jejunal feeding with early gastric feeding in critically ill patients. Crit Care Med. 2002 Apr;30(4):796-800. doi: 10.1097/00003246-200204000-00013. PMID 11940748
- [Background] Muscedere J, Dodek P, Keenan S, Fowler R, Cook D, Heyland D; VAP Guidelines Committee and the Canadian Critical Care Trials Group. Comprehensive evidence-based clinical practice guidelines for ventilator-associated pneumonia: prevention. J Crit Care. 2008 Mar;23(1):126-37. doi: 10.1016/j.jcrc.2007.11.014. PMID 18359430
- [Background] Neumann DA, DeLegge MH. Gastric versus small-bowel tube feeding in the intensive care unit: a prospective comparison of efficacy. Crit Care Med. 2002 Jul;30(7):1436-8. doi: 10.1097/00003246-200207000-00006. PMID 12130958
- [Background] Niv E, Fireman Z, Vaisman N. Post-pyloric feeding. World J Gastroenterol. 2009 Mar 21;15(11):1281-8. doi: 10.3748/wjg.15.1281. PMID 19294757
- [Background] Scolapio JS. Decreasing aspiration risk with enteral feeding. Gastrointest Endosc Clin N Am. 2007 Oct;17(4):711-6. doi: 10.1016/j.giec.2007.07.013. PMID 17967376
- [Background] Teague WG. Noninvasive ventilation in the pediatric intensive care unit for children with acute respiratory failure. Pediatr Pulmonol. 2003 Jun;35(6):418-26. doi: 10.1002/ppul.10281. PMID 12746937
- [Background] Teague WG. Non-invasive positive pressure ventilation: current status in paediatric patients. Paediatr Respir Rev. 2005 Mar;6(1):52-60. doi: 10.1016/j.prrv.2004.11.014. PMID 15698817
- [Background] Thurley PD, Hopper MA, Jobling JC, Teahon K. Fluoroscopic insertion of post-pyloric feeding tubes: success rates and complications. Clin Radiol. 2008 May;63(5):543-8. doi: 10.1016/j.crad.2007.11.005. Epub 2008 Feb 6. PMID 18374718
- [Background] Wernerman J. Intensive care unit nutrition -- nonsense or neglect? Crit Care. 2005 Jun;9(3):251-2. doi: 10.1186/cc3530. Epub 2005 Apr 20. PMID 15987414
- [Background] White H, Sosnowski K, Tran K, Reeves A, Jones M. A randomised controlled comparison of early post-pyloric versus early gastric feeding to meet nutritional targets in ventilated intensive care patients. Crit Care. 2009;13(6):R187. doi: 10.1186/cc8181. Epub 2009 Nov 25. PMID 19930728